CLINICAL TRIAL: NCT02612376
Title: Rocky Mountain Alzheimer's Disease Center at the University of Colorado School of Medicine (RMADC at UCSOM) Longitudinal Biomarker and Clinical Phenotyping Study
Brief Title: Rocky Mountain Alzheimer's Disease Center Longitudinal Biomarker and Clinical Phenotyping Study
Status: Terminated | Type: Observational
Why Stopped: Loss of funding
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1774
Record Dates: First submitted 2015-11-13; First posted 2015-11-23 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Down Syndrome; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Down Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Biospecimen Retention: Samples With DNA — Biospecimens of blood and cerebral spinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AD, DS, Mild Cognitive Impairment: Persons with age-related Mild Cognitive Impairment (MCI) or Alzheimer Disease (AD) according to clinical diagnosis, consistent with Alzheimer's Association (AA) and the National Institute on Aging (NIA) diagnostic criteria.
- Healthy Controls: * Community-dwelling controls
  * An Informant (study partner) available to complete functional interviews/survey measures annually.

SUMMARY:
This study plans to establish a large bank of blood, cerebral spinal fluid (CSF), imaging, and clinical data. These data and samples will be used for future research into the causes of Alzheimer's disease (AD), Down Syndrome (DS) and other diseases that cause thinking and memory problems. This future research will also study how treatments for these diseases work. This research may help develop new treatments for some diseases of the nervous system and help understand these diseases better.

ELIGIBILITY:
Inclusion Criteria:

1. Persons with age-related MCI or AD according to clinical diagnosis, consistent with NIA-AA diagnostic criteria
2. Community-dwelling controls, Age > 60 years
3. Ability to complete baseline assessments
4. Has an informant (study partner) available to complete functional interviews/survey measures annually

Exclusion Criteria:

* Presence of concomitant medical, neurological, or psychiatric illness or condition that in the opinion of the investigators would confound interpretation of study results. These include: Korsakoff encephalopathy; active substance abuse; hepatitis C; opportunistic brain infection; brain tumor; active neoplastic disease (skin tumors other than melanoma are not exclusionary; participants with stable prostate cancer may be included at the discretion of the project director); multiple sclerosis; history of clinically significant stroke; current evidence or history in the past 2 years of focal brain lesion, head injury with loss of consciousness, or DSM-V criteria for any major psychiatric disorder, including psychosis, major depression, bipolar disorder, alcohol or substance abuse; blindness, deafness or any other disability which may prevent the participant from participating or cooperating in the protocol.
* Presence of contraindication for MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants with Mild Cognitive Impairment (MCI), AD, healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-02; Primary Completion 2025-04 (Actual); Study Completion 2025-05 (Actual)

PRIMARY OUTCOMES:
Longitudinal collection of biospecimens and data from participants with MCI, AD, DS, healthy controls, and parents of DS individuals. | Annually for 15 years or death
  Whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Brianne M Bettcher, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No